CLINICAL TRIAL: NCT03567109
Title: Body Schema Alterations in Patients Suffering From Musculoskeletal Disorders. Does Disorder Laterality Influence Recruitment of Cerebral Areas Involved in Voluntary Motricity?
Brief Title: Body Schema Alterations in Musculoskeletal Disorders : Effect of Laterality
Acronym: Schem-TMS
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2018-A00354-51
Record Dates: First submitted 2018-06-06; First posted 2018-06-25 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Musculoskeletal Disorder; Rotator Cuff Tendinitis; Chronic Low Back Pain; Carpal Tunnel Syndrome
MeSH Terms: conditions — Musculoskeletal Diseases; Rotator Cuff Injuries; Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Shoulder rotator cuff tendinopathy: unilateral rotator cuff tendinopathy, 3 months or more duration, confirmed by imagery,
  Interventions: Other: hand laterality judgment task
- chronic low back pain: non specific chronic (3 months) low back pain
  Interventions: Other: hand laterality judgment task
- carpal tunnel syndrome: unilateral carpal tunnel syndrome, confirmed by electromyogram, 3 months or more duration
  Interventions: Other: hand laterality judgment task
- control: healthy subjects
  Interventions: Other: hand laterality judgment task

INTERVENTIONS:
Other: hand laterality judgment task — participants are asked to identify laterality of the hand presented on the screen

SUMMARY:
This study assess ocular movements in a hand laterality judgment task in a population of musculoskeletal disorders. Reaction time, error rate and visual strategy are compared between musculoskeletal disorders and healthy patients, and between the different locations of the disorder.

DETAILED DESCRIPTION:
Musculoskeletal disorders are a major public health issue. Recent studies showed that body schema alterations are involved in the chronification of those disorders. Those alterations bring the opportunity for new exploration or therapeutic solutions. Our hypothesis is that musculoskeletal disorders lead to motor imagery alterations relative to body schema disorders. Reaction time extension et error rate increase in a hand laterality judgment task would confirm that hypothesis. It is assumed that body schema alterations of patients suffering from musculoskeletal disorders could change with localisation, dependant on disorder's laterality and distality.

It is a monocentric, prospective, case-control trial, with 4 subgroups of 30 patients : shoulder rotator cuff tendinopathy, carpal tunnel syndrome, chronic low back pain, healthy subjects. We compare reaction time and error rate on a hand laterality judgement task. In that task, participants are asked to identify hand right or left laterality, when those hand is presented on a computer screen, by answering with the keyboard. Hands are shown on palmar or dorsal view and with 12 different angles of rotation. An eye-tracking device register participant eye movements during the task.

ELIGIBILITY:
Inclusion Criteria:

* normal visual acuity
* social security affiliation
* signing consent
* rotator cuff tendinopathy, chronic low back pain, carpal tunnel syndrome or healthy subject

Exclusion Criteria:

* recent trauma or surgery
* psychiatric or neurological disorder
* psychotropic consumption
* previous experience with motor imagery
* bad french comprehension
* protected persons
* other painful affection than the inclusion criteria

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients refered to the Hospital University of Angers or the Hand Center in Trelazé for one of the musculoskeletal disorders meeting the inclusion criterias.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
error rate at the hand laterality judgment task | 1 hour
  number of errors divided by the total number of hands presented
reaction time | 1 hour
  time to press on the keyboard the answer "Right" or "Left" after the hand was presented

SECONDARY OUTCOMES:
visual strategy | 1 hour
  assessment of the image's areas most fixed with the eyes

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: Undecided